CLINICAL TRIAL: NCT01620528
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Elagolix in Subjects With Moderate to Severe Endometriosis-Associated Pain
Brief Title: A Clinical Study to Evaluate the Safety and Efficacy of Elagolix in Subjects With Moderate to Severe Endometriosis-Associated Pain
Acronym: ELARIS EM-I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M12-665
Record Dates: First submitted 2012-05-15; First posted 2012-06-15 (Estimated); Results first posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2017-03

CONDITIONS: Endometriosis
Keywords: Gonadotropin-Releasing Hormone Antagonist; Endometriosis associated pain; Dysmenorrhea (DYS); Non-Menstrual Pelvic Pain (NMPP); Elagolix
MeSH Terms: conditions — Endometriosis; Dysmenorrhea | interventions — elagolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Elagolix 150 mg QD (Experimental): Elagolix 150 mg once daily (QD) for the 6-month Treatment Period
  Interventions: Drug: elagolix
- Elagolix 200 mg BID (Experimental): Elagolix 200 mg twice daily (BID) for the 6-month Treatment Period
  Interventions: Drug: elagolix
- Placebo (Placebo Comparator): Placebo BID for the 6-month Treatment Period
  Interventions: Other: placebo

INTERVENTIONS:
Drug: elagolix — oral tablet
  Other Names: ABT-620, elagolix sodium
  Arms: Elagolix 150 mg QD; Elagolix 200 mg BID
Other: placebo — oral tablet
  Arms: Placebo

SUMMARY:
A randomized study evaluating the safety and efficacy of elagolix in the management of moderate to severe endometriosis-associated pain in adult premenopausal female participants.

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, double-blind, placebo-controlled, randomized study to assess the safety and efficacy of two doses of elagolix versus placebo in premenopausal 18 to 49 year old women with moderate to severe endometriosis-associated pain. The study consists of 4 periods: 1) Washout Period (if applicable); 2) a Screening Period of up to 100 days prior to first dose; 3) a 6 month Treatment Period; and 4) a Post treatment Follow-up Period of up to 12 months (if applicable). An electronic diary will be dispensed and training provided to record endometriosis-associated pain, uterine bleeding, and analgesic medication use for endometriosis-associated pain on a daily basis. Pregnancy testing will be performed monthly throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal female, between 18 and 49 years of age, inclusive, at the time of signing consent.
2. Clinical diagnosis of endometriosis (laparoscopy or laparotomy) performed within 10 years of entry into Washout (if applicable) or Screening.
3. Agrees to use required birth control methods during the entire length of participation in the study.
4. Subject has a Composite Pelvic Signs and Symptoms Score total score of ≥ 6 at Screening with a score of at least 2 for dysmenorrhea AND at least 2 for non-menstrual pelvic pain. 5. Subjects must have at least two menstrual cycles 24 to 38 days within the Screening Period, prior to Day 1

Exclusion Criteria:

1. Subject is pregnant or breast feeding or is planning a pregnancy within the next 24 months or is less than 6 months postpartum, post-abortion, or post-pregnancy at the time of entry into the Screening Period.
2. Subject has a history of previous non-response to Gonadotropin-releasing hormone (GnRH) agonists, GnRH antagonists, Depot Medroxyprogesterone Acetate, or aromatase inhibitors as assessed by subject report of no improvement in dysmenorrhea or non-menstrual pelvic pain (subject report of partial response to or side effects from these agents is not exclusionary).
3. Subject has chronic pelvic pain that is not caused by endometriosis that requires chronic analgesic or other chronic therapy, or that would interfere with the assessment of endometriosis related pain.
4. Clinically significant gynecologic condition identified on Screening transvaginal ultrasound or endometrial biopsy.
5. Subject has a history of osteoporosis or other metabolic bone disease.
6. Subject has a current history of undiagnosed abnormal genital bleeding.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 872 (Actual)
Dates: Start 2012-05-22; Primary Completion 2014-11-14 (Actual); Study Completion 2015-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Duan, MD, Study Director — AbbVie

REFERENCES:
- [Result] Taylor HS, Giudice LC, Lessey BA, Abrao MS, Kotarski J, Archer DF, Diamond MP, Surrey E, Johnson NP, Watts NB, Gallagher JC, Simon JA, Carr BR, Dmowski WP, Leyland N, Rowan JP, Duan WR, Ng J, Schwefel B, Thomas JW, Jain RI, Chwalisz K. Treatment of Endometriosis-Associated Pain with Elagolix, an Oral GnRH Antagonist. N Engl J Med. 2017 Jul 6;377(1):28-40. doi: 10.1056/NEJMoa1700089. Epub 2017 May 19. PMID 28525302
- [Derived] Beck D, Winzenborg I, Liu M, Degner J, Mostafa NM, Noertersheuser P, Shebley M. Population Pharmacokinetics of Elagolix in Combination with Low-Dose Estradiol/Norethindrone Acetate in Women with Uterine Fibroids. Clin Pharmacokinet. 2022 Apr;61(4):577-587. doi: 10.1007/s40262-021-01096-w. Epub 2021 Dec 8. PMID 34878624
- [Derived] Abrao MS, Surrey E, Gordon K, Snabes MC, Wang H, Ijacu H, Taylor HS. Reductions in endometriosis-associated pain among women treated with elagolix are consistent across a range of baseline characteristics reflective of real-world patients. BMC Womens Health. 2021 Jun 16;21(1):246. doi: 10.1186/s12905-021-01385-3. PMID 34134684
- [Derived] Stodtmann S, Nader A, Polepally AR, Suleiman AA, Winzenborg I, Noertersheuser P, Ng J, Mostafa NM, Shebley M. Validation of a quantitative systems pharmacology model of calcium homeostasis using elagolix Phase 3 clinical trial data in women with endometriosis. Clin Transl Sci. 2021 Jul;14(4):1611-1619. doi: 10.1111/cts.13040. Epub 2021 May 7. PMID 33963686
- [Derived] Beck D, Winzenborg I, Gao W, Mostafa NM, Noertersheuser P, Chiuve SE, Owens C, Shebley M. Integrating real-world data and modeling to project changes in femoral neck bone mineral density and fracture risk in premenopausal women. Clin Transl Sci. 2021 Jul;14(4):1452-1463. doi: 10.1111/cts.13006. Epub 2021 Apr 8. PMID 33650259
- [Derived] Agarwal SK, Singh SS, Archer DF, Mai Y, Chwalisz K, Gordon K, Surrey E. Endometriosis-Related Pain Reduction During Bleeding and Nonbleeding Days in Women Treated with Elagolix. J Pain Res. 2021 Feb 2;14:263-271. doi: 10.2147/JPR.S284703. eCollection 2021. PMID 33564263
- [Derived] Pokrzywinski RM, Soliman AM, Snabes MC, Chen J, Taylor HS, Coyne KS. Responsiveness and thresholds for clinically meaningful changes in worst pain numerical rating scale for dysmenorrhea and nonmenstrual pelvic pain in women with moderate to severe endometriosis. Fertil Steril. 2021 Feb;115(2):423-430. doi: 10.1016/j.fertnstert.2020.07.013. Epub 2020 Oct 14. PMID 33066973
- [Derived] Abbas Suleiman A, Nader A, Winzenborg I, Beck D, Polepally AR, Ng J, Noertersheuser P, Mostafa NM. Exposure-Safety Analyses Identify Predictors of Change in Bone Mineral Density and Support Elagolix Labeling for Endometriosis-Associated Pain. CPT Pharmacometrics Syst Pharmacol. 2020 Nov;9(11):639-648. doi: 10.1002/psp4.12560. Epub 2020 Oct 8. PMID 32945631
- [Derived] Taylor HS, Soliman AM, Johns B, Pokrzywinski RM, Snabes M, Coyne KS. Health-Related Quality of Life Improvements in Patients With Endometriosis Treated With Elagolix. Obstet Gynecol. 2020 Sep;136(3):501-509. doi: 10.1097/AOG.0000000000003917. PMID 32769633
- [Derived] Winzenborg I, Polepally AR, Nader A, Mostafa NM, Noertersheuser P, Ng J. Effect of Elagolix Exposure on Clinical Efficacy End Points in Phase III Trials in Women With Endometriosis-Associated Pain: An Application of Markov Model. CPT Pharmacometrics Syst Pharmacol. 2020 Aug;9(8):466-475. doi: 10.1002/psp4.12545. Epub 2020 Jul 31. PMID 32621325
- [Derived] Surrey ES, Soliman AM, Palac HL, Agarwal SK. Impact of Elagolix on Workplace and Household Productivity Among Women with Moderate to Severe Pain Associated with Endometriosis: A Pooled Analysis of Two Phase III Trials. Patient. 2019 Dec;12(6):651-660. doi: 10.1007/s40271-019-00394-7. PMID 31654294
- [Derived] Pokrzywinski RM, Soliman AM, Chen J, Snabes M, Diamond MP, Surrey E, Coyne KS. Impact of elagolix on work loss due to endometriosis-associated pain: estimates based on the results of two phase III clinical trials. Fertil Steril. 2019 Sep;112(3):545-551. doi: 10.1016/j.fertnstert.2019.04.031. Epub 2019 Jun 18. PMID 31227284
- [Derived] Surrey ES, Soliman AM, Agarwal SK, Snabes MC, Diamond MP. Impact of elagolix treatment on fatigue experienced by women with moderate to severe pain associated with endometriosis. Fertil Steril. 2019 Aug;112(2):298-304.e3. doi: 10.1016/j.fertnstert.2019.02.031. Epub 2019 Apr 13. PMID 30992150
- [Derived] Wang ST, Johnson SJ, Mitchell D, Soliman AM, Vora JB, Agarwal SK. Cost-effectiveness of elagolix versus leuprolide acetate for treating moderate-to-severe endometriosis pain in the USA. J Comp Eff Res. 2019 Apr;8(5):337-355. doi: 10.2217/cer-2018-0124. Epub 2019 Feb 6. PMID 30724096
- [Derived] Winzenborg I, Nader A, Polepally AR, Liu M, Degner J, Klein CE, Mostafa NM, Noertersheuser P, Ng J. Population Pharmacokinetics of Elagolix in Healthy Women and Women with Endometriosis. Clin Pharmacokinet. 2018 Oct;57(10):1295-1306. doi: 10.1007/s40262-018-0629-6. PMID 29476499

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After completing the Treatment Period, participants (who were eligible and provided consent) entered a separate continuous-use extension study (Study M12-667, NCT01760954).
Pre-assignment Details: Participants who prematurely discontinued from study drug and those who declined to participate in or who did not qualify for the continuous-use extension study, except for those who became pregnant, could elect to enter the Post-Treatment Follow-Up (PTFU) Period within this study for up to 12 additional months.
Groups:
- Placebo: Placebo twice daily (BID) for the 6-month Treatment Period
- Elagolix 200 mg BID: Elagolix 200 mg BID for the 6-month Treatment Period
Period: Treatment Period
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Started | 374 | 249 | 249 (1 subject did not receive study drug)
Completed | 274 | 196 | 183
Not Completed | 100 | 53 | 66
Not completed — Did Not Receive Study Drug | 0 | 0 | 1
Not completed — Withdrawal by Subject | 35 | 21 | 16
Not completed — Adverse Event | 17 | 13 | 21
Not completed — Lost to Follow-up | 16 | 8 | 14
Not completed — Other | 9 | 5 | 7
Not completed — Subject Noncompliant | 11 | 2 | 2
Not completed — Pregnancy | 7 | 2 | 2
Not completed — Surgery/Invasive Intervention | 5 | 1 | 3
Not completed — Exclusionary Medication Received | 0 | 1 | 0
Period: Post-Treatment Follow-Up Period
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Started | 68 (elected to enter the PTFU Period) | 48 (elected to enter the PTFU Period) | 51 (elected to enter the PTFU Period)
Completed PTFU Month 6 (Met criteria (reported post-treatment menses, met the DXA criteria, and had a PTFU Month 6 visit).) | 46 | 26 (Met criteria (reported a post-treatment menses, met the DXA criteria, and had a PTFU Month 6 visit).) | 18 (Met criteria (reported a post-treatment menses, met the DXA criteria, and had a PTFU Month 6 visit).)
Completed PTFU Month 12 | 2 | 5 | 19
Completed | 48 | 31 | 37
Not Completed | 20 | 17 | 14
Not completed — Withdrawal by Subject | 3 | 7 | 3
Not completed — Lost to Follow-up | 3 | 2 | 4
Not completed — Exclusionary Medication Received | 0 | 1 | 1
Not completed — Surgery/Invasive Intervention | 8 | 3 | 4
Not completed — Other | 6 | 4 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug
Groups:
- Elagolix 150 mg QD: Elagolix 150 mg QD for the 6-month Treatment Period
- Total: Total of all reporting groups
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID | Total
Number analyzed (Participants) | 374 | 249 | 248 | 871
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (6.35) | 31.5 (5.99) | 31.2 (6.33) | 31.5 (6.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 374 | 249 | 248 | 871
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders at Month 3 Based on Daily Assessment of Dysmenorrhea (DYS)
Description: The DYS pain scale ranges from 0 (none) to 3 (severe). The criteria for a responder was based on a pre-defined threshold and accounted for analgesic use.
Time Frame: At Month 3 of the Treatment Period
Population: The modified intent-to-treat (mITT) analysis set; all randomized participants who took at least 1 dose of randomized, double-blind study drug. Population included mITT participants who either had data during the Month 3 35-day window or who prematurely discontinued prior to or at Month 3 and met the rules for last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 373 | 248 | 244
percentage of participants | 19.6 | 46.4 | 75.8
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, Regression, Logistic

2. Primary Outcome: Percentage of Responders at Month 3 Based on Daily Assessment of Non-Menstrual Pelvic Pain (NMPP)
Description: The NMPP pain scale ranges from 0 (none) to 3 (severe). The criteria for a responder was based on a pre-defined threshold and accounted for analgesic use.
Time Frame: At Month 3 of Treatment Period
Population: The mITT analysis set; all randomized participants who took at least 1 dose of randomized, double-blind study drug. Population included mITT participants who either had data during the Month 3 35-day window or who prematurely discontinued prior to or at Month 3 and met the rules for last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 373 | 248 | 244
percentage of participants | 36.5 | 50.4 | 54.5
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, Regression, Logistic

3. Secondary Outcome: Change From Baseline to Month 3 in Numeric Rating Scale (NRS) Scores
Description: The NRS for overall endometriosis-associated pain ranges 0 (none) to 10 (worst pain ever).
Time Frame: Baseline, Month 3 of the Treatment Period
Population: The mITT analysis set included all randomized participants who took at least 1 dose of randomized, double-blind study drug. Observed cases.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 329 | 226 | 213
units on a scale | -1.09 (0.098) | -1.74 (0.120) | -2.39 (0.122)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Ranked secondary efficacy endpoint 1 of 7; Test type: Superiority; p < 0.001, mixed-effects model; Difference in LS Mean Change = -0.65, Standard Error of Mean 0.155
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Ranked secondary efficacy endpoint 1 of 7; Test type: Superiority; p < 0.001, mixed-effects model; Difference in LS Mean Change = -1.30, Standard Error of Mean 0.156

4. Secondary Outcome: Change From Baseline to Month 6 in DYS
Description: The DYS pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 6 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 288 | 198 | 182
units on a scale | -0.44 (0.047) | -0.89 (0.057) | -1.75 (0.059)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Ranked secondary efficacy endpoint 2 of 7; Test type: Superiority; p < 0.001, mixed-effects model; Difference in LS Mean Change = -0.45, Standard Error of Mean 0.074
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Ranked secondary efficacy endpoint 2 of 7; Test type: Superiority; p < 0.001, mixed-effects model; Difference in Least Squares Mean = -1.32, Standard Error of Mean 0.076

5. Secondary Outcome: Change From Baseline to Month 6 in NMPP
Description: The NMPP pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 6 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 288 | 198 | 182
units on a scale | -0.31 (0.035) | -0.48 (0.043) | -0.72 (0.044)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Ranked secondary efficacy endpoint 3 of 7; Test type: Superiority; p = 0.004, mixed-effects model; Difference in LS Mean Change = -0.16, Standard Error of Mean 0.056
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Ranked secondary efficacy endpoint 3 of 7; Test type: Superiority; p < 0.001, mixed-effects model; Least Squares Mean Difference = -0.41, Standard Error of Mean 0.057

6. Secondary Outcome: Change From Baseline to Month 3 in Analgesic Use Across Both Classes of Rescue Analgesics
Description: Permitted rescue medications included the nonsteroidal anti-inflammatory drug naproxen (500 mg), the narcotic analgesics 5 mg hydrocodone + 300 or 325 mg acetaminophen, and 30 mg codeine + 300 mg acetaminophen. Assessment was based on average pill counts.
Time Frame: Baseline, Month 3 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: pills
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 329 | 226 | 213
pills | -0.29 (0.032) | -0.29 (0.039) | -0.55 (0.040)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Ranked secondary efficacy endpoint 4 of 7; Test type: Superiority; p = 0.910, mixed-effects model; Difference in LS Mean Change = -0.01, Standard Error of Mean 0.051
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Ranked secondary efficacy endpoint 4 of 7; Test type: Superiority; p < 0.001, mixed-effects model; Difference in LS Mean Change = -0.26, Standard Error of Mean 0.051

7. Secondary Outcome: Change From Baseline to Month 6 in Analgesic Use Across Both Classes of Rescue Analgesics
Description: Permitted rescue medications included the nonsteroidal anti-inflammatory drug naproxen (500 mg), the narcotic analgesics 5 mg hydrocodone + 300 or 325 mg acetaminophen and 30 mg codeine + 300 mg acetaminophen. Assessment was based on average pill counts.
Time Frame: Baseline, Month 6 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: pills
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 288 | 198 | 182
pills | -0.27 (0.036) | -0.35 (0.043) | -0.56 (0.045)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Ranked secondary efficacy endpoint 5 of 7; Test type: Superiority; p = 0.185, mixed-effects model; Difference in LS Mean Change = -0.07, Standard Error of Mean 0.056
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Ranked secondary efficacy endpoint 5 of 7; Test type: Superiority; p < 0.001, mixed-effects model; Least Squares Mean Difference = -0.28, Standard Error of Mean 0.057

8. Secondary Outcome: Change From Baseline to Month 3 in Dyspareunia (DYSP)
Description: The DYSP pain scale ranges from 0 (absent) to 3 (severe).
Time Frame: Baseline, Month 3 of Treatment Period
Population: The mITT analysis set included all randomized participants who took at least 1 dose of randomized, double-blind study drug. Observed cases. Participants who responded "not applicable" for the entire time point and at Baseline are excluded from the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 246 | 171 | 153
units on a scale | -0.29 (0.041) | -0.39 (0.050) | -0.49 (0.052)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Ranked secondary efficacy endpoint 6 of 7; Test type: Superiority; p = 0.144, mixed-effects model; Difference in LS Mean Change = -0.09, Standard Error of Mean 0.065
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Ranked secondary efficacy endpoint 6 of 7; Test type: Superiority; p = 0.003, mixed-effects model; Difference in LS Mean Change = -0.20, Standard Error of Mean 0.067

9. Secondary Outcome: Change From Baseline to Month 3 in Use of Narcotic Class of Medication (Opioids)
Description: Permitted rescue narcotic analgesics included 5 mg hydrocodone + 300 or 325 mg acetaminophen and 30 mg codeine + 300 mg acetaminophen. Assessment was based on average pill counts.
Time Frame: Baseline, Month 3 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: pills
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 329 | 226 | 213
pills | -0.10 (0.024) | -0.07 (0.029) | -0.22 (0.029)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Ranked secondary efficacy endpoint 7 of 7; Test type: Superiority; p = 0.424, mixed-effects model; Difference in LS Mean Change = 0.03, Standard Error of Mean 0.037
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Ranked secondary efficacy endpoint 7 of 7; Test type: Superiority; p = 0.002, mixed-effects model; Difference in LS Mean Change = -0.12, Standard Error of Mean 0.038

10. Secondary Outcome: Percentage of Responders at Month 1 Based on Daily Assessment of DYS
Description: as for outcome 1
Time Frame: At Month 1 of the Treatment Period
Population: The mITT analysis set included all randomized participants who took at least 1 dose of randomized, double-blind study drug. Last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 372 | 248 | 245
percentage of participants | 14.5 | 35.1 | 44.1
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, Regression, Logistic

11. Secondary Outcome: Percentage of Responders at Month 2 Based on Daily Assessment of DYS
Description: as for outcome 1
Time Frame: At Month 2 of the Treatment Period
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 373 | 248 | 244
percentage of participants | 17.2 | 44.8 | 71.3
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, Regression, Logistic

12. Secondary Outcome: Percentage of Responders at Month 4 Based on Daily Assessment of DYS
Description: as for outcome 1
Time Frame: At Month 4 of the Treatment Period
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 373 | 248 | 243
percentage of participants | 21.7 | 47.6 | 75.3
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, Regression, Logistic

13. Secondary Outcome: Percentage of Responders at Month 5 Based on Daily Assessment of DYS
Description: as for outcome 1
Time Frame: At Month 5 of the Treatment Period
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 371 | 247 | 243
percentage of participants | 24.3 | 45.7 | 79.0
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, Regression, Logistic

14. Secondary Outcome: Percentage of Responders at Month 6 Based on Daily Assessment of DYS
Description: as for outcome 1
Time Frame: At Month 6 of the Treatment Period
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 372 | 247 | 243
percentage of participants | 23.1 | 42.1 | 75.3
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, Regression, Logistic

15. Secondary Outcome: Percentage of Responders at Month 1 Based on Daily Assessment of NMPP
Description: as for outcome 2
Time Frame: At Month 1 of Treatment Period
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 372 | 248 | 245
percentage of participants | 25.8 | 32.3 | 33.9
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.103, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p = 0.023, Regression, Logistic

16. Secondary Outcome: Percentage of Responders at Month 2 Based on Daily Assessment of NMPP
Description: as for outcome 2
Time Frame: At Month 2 of Treatment Period
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 373 | 248 | 244
percentage of participants | 32.2 | 41.1 | 46.3
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.031, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, Regression, Logistic

17. Secondary Outcome: Percentage of Responders at Month 4 Based on Daily Assessment of NMPP
Description: as for outcome 2
Time Frame: At Month 4 of Treatment Period
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 373 | 248 | 243
percentage of participants | 35.4 | 53.2 | 63.8
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, Regression, Logistic

18. Secondary Outcome: Percentage of Responders at Month 5 Based on Daily Assessment of NMPP
Description: as for outcome 2
Time Frame: At Month 5 of Treatment Period
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 371 | 247 | 243
percentage of participants | 38.3 | 49.8 | 62.1
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.005, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, Regression, Logistic

19. Secondary Outcome: Percentage of Responders at Month 6 Based on Daily Assessment of NMPP
Description: as for outcome 2
Time Frame: At Month 6 of Treatment Period
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 372 | 247 | 243
percentage of participants | 34.9 | 45.7 | 62.1
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.008, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, Regression, Logistic

20. Secondary Outcome: Percentage of Responders at Month 1 for DYSP
Description: The DYSP pain scale ranged from 0 (absent) to 3 (severe). The criteria for a responder was based on a pre-defined threshold and accounted for analgesic use.
Time Frame: At Month 1 of the Treatment Period
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 293 | 191 | 176
percentage of participants | 26.3 | 30.4 | 31.8
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.306, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p = 0.239, Regression, Logistic

21. Secondary Outcome: Percentage of Responders at Month 2 for DYSP
Description: as for outcome 20
Time Frame: At Month 2 of the Treatment Period
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 287 | 190 | 179
percentage of participants | 33.1 | 33.7 | 44.7
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.855, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p = 0.012, Regression, Logistic

22. Secondary Outcome: Percentage of Responders at Month 4 for DYSP
Description: as for outcome 20
Time Frame: At Month 4 of the Treatment Period
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 278 | 185 | 168
percentage of participants | 33.1 | 44.3 | 54.2
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.010, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, Regression, Logistic

23. Secondary Outcome: Percentage of Responders at Month 5 for DYSP
Description: as for outcome 20
Time Frame: At Month 5 of the Treatment Period
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 275 | 183 | 166
percentage of participants | 35.3 | 43.7 | 54.8
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.061, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, Regression, Logistic

24. Secondary Outcome: Percentage of Responders at Month 6 for DYSP
Description: as for outcome 20
Time Frame: At Month 6 of the Treatment Period
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 270 | 187 | 161
percentage of participants | 33.3 | 39.6 | 50.3
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.126, Regression, Logistic
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, Regression, Logistic

25. Secondary Outcome: Change From Baseline to Month 1 in Mean Pain Score for DYS
Description: The DYS pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 1 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 372 | 248 | 245
units on a scale | -0.33 (0.044) | -0.83 (0.054) | -0.98 (0.054)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.50, 97.5% CI 2-sided [-0.65 to -0.34], Standard Error of Mean 0.070
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.65, 97.5% CI 2-sided [-0.81 to -0.49], Standard Error of Mean 0.070

26. Secondary Outcome: Change From Baseline to Month 2 in Mean Pain Score for DYS
Description: The DYS pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 2 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 348 | 232 | 221
units on a scale | -0.32 (0.042) | -0.96 (0.052) | -1.68 (0.053)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.64, 97.5% CI 2-sided [-0.79 to -0.49], Standard Error of Mean 0.067
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -1.36, 97.5% CI 2-sided [-1.51 to -1.20], Standard Error of Mean 0.068

27. Secondary Outcome: Change From Baseline to Month 3 in Mean Pain Score for DYS
Description: The DYS pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 3 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 329 | 226 | 213
units on a scale | -0.35 (0.043) | -1.03 (0.052) | -1.73 (0.054)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.68, 97.5% CI 2-sided [-0.83 to -0.53], Standard Error of Mean 0.068
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -1.39, 97.5% CI 2-sided [-1.54 to -1.23], Standard Error of Mean 0.069

28. Secondary Outcome: Change From Baseline to Month 4 in Mean Pain Score for DYS
Description: The DYS pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 4 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 316 | 219 | 198
units on a scale | -0.40 (0.045) | -1.05 (0.054) | -1.72 (0.057)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.65, 97.5% CI 2-sided [-0.81 to -0.49], Standard Error of Mean 0.071
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -1.32, 97.5% CI 2-sided [-1.49 to -1.16], Standard Error of Mean 0.072

29. Secondary Outcome: Change From Baseline to Month 5 in Mean Pain Score for DYS
Description: The DYS pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 5 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 299 | 202 | 191
units on a scale | -0.43 (0.045) | -1.02 (0.054) | -1.84 (0.056)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.59, 97.5% CI 2-sided [-0.75 to -0.43], Standard Error of Mean 0.071
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -1.41, 97.5% CI 2-sided [-1.58 to -1.25], Standard Error of Mean 0.072

30. Secondary Outcome: Percent Change From Baseline to Month 1 in Mean Pain Score for DYS
Description: The DYS pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 1 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 372 | 248 | 245
percentage change | -14.35 (2.079) | -38.42 (2.547) | -45.35 (2.562)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -24.07, 97.5% CI 2-sided [-31.45 to -16.69], Standard Error of Mean 3.288
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -31.01, 97.5% CI 2-sided [-38.41 to -23.60], Standard Error of Mean 3.299

31. Secondary Outcome: Percent Change From Baseline to Month 2 in Mean Pain Score for DYS
Description: The DYS pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 2 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 348 | 232 | 221
percentage change | -13.44 (1.965) | -44.23 (2.407) | -77.22 (2.460)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = -30.79, mixed-effects model; LS Mean of Difference = -30.79, 97.5% CI 2-sided [-37.77 to -23.82], Standard Error of Mean 3.107
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -63.78, 97.5% CI 2-sided [-70.85 to -56.71], Standard Error of Mean 3.148

32. Secondary Outcome: Percent Change From Baseline to Month 3 in Mean Pain Score for DYS
Description: The DYS pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 3 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 329 | 226 | 213
percentage change | -14.80 (2.022) | -47.01 (2.451) | -79.74 (2.519)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -32.21, 97.5% CI 2-sided [-39.35 to -25.08], Standard Error of Mean 3.177
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -64.94, 97.5% CI 2-sided [-72.19 to -57.68], Standard Error of Mean 3.230

33. Secondary Outcome: Percent Change From Baseline to Month 4 in Mean Pain Score for DYS
Description: The DYS pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 4 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 316 | 219 | 198
percentage change | -18.08 (2.088) | -48.02 (2.519) | -79.98 (2.627)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -29.94, 97.5% CI 2-sided [-37.28 to -22.59], Standard Error of Mean 3.272
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -61.90, 97.5% CI 2-sided [-69.44 to -54.36], Standard Error of Mean 3.356

34. Secondary Outcome: Percent Change From Baseline to Month 5 in Mean Pain Score for DYS
Description: The DYS pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 5 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 299 | 202 | 191
percentage change | -18.09 (2.072) | -46.72 (2.517) | -84.58 (2.595)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -28.63, 97.5% CI 2-sided [-35.96 to -21.31], Standard Error of Mean 3.260
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -66.50, 97.5% CI 2-sided [-73.95 to -59.04], Standard Error of Mean 3.321

35. Secondary Outcome: Percent Change From Baseline to Month 6 in Mean Pain Score for DYS
Description: The DYS pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 6 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 288 | 198 | 182
percentage change | -19.21 (2.217) | -40.60 (2.681) | -79.99 (2.782)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -21.39, 97.5% CI 2-sided [-29.20 to -13.57], Standard Error of Mean 3.479
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -60.78, 97.5% CI 2-sided [-68.77 to -52.79], Standard Error of Mean 3.557

36. Secondary Outcome: Change From Baseline to Month 1 in Mean Pain Score for NMPP
Description: The NMPP pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 1 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 372 | 248 | 245
units on a scale | -0.16 (0.023) | -0.22 (0.028) | -0.26 (0.028)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.111, mixed-effects model; LS Mean of Difference = -0.06, 97.5% CI 2-sided [-0.14 to 0.02], Standard Error of Mean 0.036
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p = 0.008, mixed-effects model; LS Mean of Difference = -0.10, 97.5% CI 2-sided [-0.18 to -0.01], Standard Error of Mean 0.036

37. Secondary Outcome: Change From Baseline to Month 2 in Mean Pain Score for NMPP
Description: The NMPP pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 2 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 348 | 232 | 221
units on a scale | -0.26 (0.028) | -0.33 (0.035) | -0.44 (0.035)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.092, mixed-effects model; LS Mean of Difference = -0.08, 97.5% CI 2-sided [-0.18 to 0.02], Standard Error of Mean 0.045
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.18, 97.5% CI 2-sided [-0.28 to -0.08], Standard Error of Mean 0.045

38. Secondary Outcome: Change From Baseline to Month 3 in Mean Pain Score for NMPP
Description: The NMPP pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 3 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 329 | 226 | 213
units on a scale | -0.32 (0.032) | -0.44 (0.039) | -0.61 (0.039)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.017, mixed-effects model; LS Mean of Difference = -0.12, 97.5% CI 2-sided [-0.23 to -0.01], Standard Error of Mean 0.050
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.29, 97.5% CI 2-sided [-0.41 to -0.18], Standard Error of Mean 0.050

39. Secondary Outcome: Change From Baseline to Month 4 in Mean Pain Score for NMPP
Description: The NMPP pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 4 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 316 | 219 | 198
units on a scale | -0.33 (0.034) | -0.51 (0.041) | -0.72 (0.042)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.19, 97.5% CI 2-sided [-0.31 to -0.07], Standard Error of Mean 0.053
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.39, 97.5% CI 2-sided [-0.51 to -0.27], Standard Error of Mean 0.054

40. Secondary Outcome: Change From Baseline to Month 5 in Mean Pain Score for NMPP
Description: The NMPP pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 5 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 299 | 202 | 191
units on a scale | -0.34 (0.034) | -0.49 (0.041) | -0.74 (0.042)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.004, mixed-effects model; LS Mean of Difference = -0.15, 97.5% CI 2-sided [-0.27 to -0.03], Standard Error of Mean 0.053
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.39, 97.5% CI 2-sided [-0.52 to -0.27], Standard Error of Mean 0.054

41. Secondary Outcome: Percent Change From Baseline to Month 1 in Mean Pain Score for NMPP
Description: The NMPP pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 1 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 372 | 248 | 245
percentage change | -7.51 (1.736) | -13.74 (2.131) | -15.23 (2.139)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.024, mixed-effects model; LS Mean of Difference = -6.23, 97.5% CI 2-sided [-12.40 to -0.06], Standard Error of Mean 2.748
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p = 0.005, mixed-effects model; LS Mean of Difference = -7.72, 97.5% CI 2-sided [-13.90 to -1.53], Standard Error of Mean 2.756

42. Secondary Outcome: Percent Change From Baseline to Month 2 in Mean Pain Score for NMPP
Description: The NMPP pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 2 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 348 | 232 | 221
percentage change | -13.81 (2.039) | -19.50 (2.501) | -27.53 (2.529)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.078, mixed-effects model; LS Mean of Difference = -5.69, 97.5% CI 2-sided [-12.93 to 1.56], Standard Error of Mean 3.226
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -13.72, 97.5% CI 2-sided [-21.01 to -6.42], Standard Error of Mean 3.249

43. Secondary Outcome: Percent Change From Baseline to Month 3 in Mean Pain Score for NMPP
Description: The NMPP pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 3 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 329 | 226 | 213
percentage change | -17.64 (2.204) | -26.10 (2.688) | -40.13 (2.737)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.015, mixed-effects model; LS Mean of Difference = -8.47, 97.5% CI 2-sided [-16.27 to -0.66], Standard Error of Mean 3.475
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -22.49, 97.5% CI 2-sided [-30.38 to -14.60], Standard Error of Mean 3.514

44. Secondary Outcome: Percent Change From Baseline to Month 4 in Mean Pain Score for NMPP
Description: The NMPP pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 4 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 316 | 219 | 198
percentage change | -17.94 (2.333) | -32.05 (2.837) | -48.35 (2.909)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -14.11, 97.5% CI 2-sided [-22.36 to -5.87], Standard Error of Mean 3.673
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -30.41, 97.5% CI 2-sided [-38.78 to -22.04], Standard Error of Mean 3.729

45. Secondary Outcome: Percent Change From Baseline to Month 5 in Mean Pain Score for NMPP
Description: The NMPP pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 5 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 299 | 202 | 191
percentage change | -19.60 (2.371) | -31.15 (2.888) | -49.28 (2.954)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.002, mixed-effects model; LS Mean of Difference = -11.55, 97.5% CI 2-sided [-19.94 to -3.16], Standard Error of Mean 3.736
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -29.68, 97.5% CI 2-sided [-38.19 to -21.18], Standard Error of Mean 3.788

46. Secondary Outcome: Percent Change From Baseline to Month 6 in Mean Pain Score for NMPP
Description: The NMPP pain scale ranges from 0 (none) to 3 (severe).
Time Frame: Baseline, Month 6 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 288 | 198 | 182
percentage change | -18.17 (2.418) | -30.55 (2.939) | -48.14 (3.019)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.001, mixed-effects model; LS Mean of Difference = -12.37, 97.5% CI 2-sided [-20.92 to -3.83], Standard Error of Mean 3.805
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -29.97, 97.5% CI 2-sided [-38.66 to -21.28], Standard Error of Mean 3.868

47. Secondary Outcome: Change From Baseline to Month 1 in Mean Pain Score of DYSP
Description: The DYSP pain scale ranged from 0 (absent) to 3 (severe).
Time Frame: Baseline, Month 1 of Treatment Period
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 293 | 191 | 176
units on a scale | -0.18 (0.032) | -0.29 (0.040) | -0.22 (0.042)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.038, mixed-effects model; LS Mean of Difference = -0.11, 97.5% CI 2-sided [-0.22 to 0.01], Standard Error of Mean 0.052
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p = 0.488, mixed-effects model; LS Mean of Difference = -0.04, 97.5% CI 2-sided [-0.16 to 0.08], Standard Error of Mean 0.053

48. Secondary Outcome: Change From Baseline to Month 2 in Mean Pain Score of DYSP
Description: The DYSP pain scale ranged from 0 (absent) to 3 (severe).
Time Frame: Baseline, Month 2 of Treatment Period
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 267 | 178 | 165
units on a scale | -0.26 (0.038) | -0.33 (0.046) | -0.38 (0.048)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.252, mixed-effects model; LS Mean of Difference = -0.07, 97.5% CI 2-sided [-0.20 to 0.07], Standard Error of Mean 0.060
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p = 0.058, mixed-effects model; LS Mean of Difference = -0.12, 97.5% CI 2-sided [-0.25 to 0.02], Standard Error of Mean 0.061

49. Secondary Outcome: Change From Baseline to Month 4 in Mean Pain Score of DYSP
Description: The DYSP pain scale ranged from 0 (absent) to 3 (severe).
Time Frame: Baseline, Month 4 of Treatment Period
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 231 | 164 | 139
units on a scale | -0.27 (0.044) | -0.45 (0.053) | -0.61 (0.056)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.009, mixed-effects model; LS Mean of Difference = -0.18, 97.5% CI 2-sided [-0.34 to -0.03], Standard Error of Mean 0.069
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.34, 97.5% CI 2-sided [-0.50 to -0.18], Standard Error of Mean 0.071

50. Secondary Outcome: Change From Baseline to Month 5 in Mean Pain Score of DYSP
Description: The DYSP pain scale ranged from 0 (absent) to 3 (severe).
Time Frame: Baseline, Month 5 of Treatment Period
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 217 | 149 | 131
units on a scale | -0.30 (0.047) | -0.44 (0.056) | -0.57 (0.060)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.060, mixed-effects model; LS Mean of Difference = -0.14, 97.5% CI 2-sided [-0.30 to 0.03], Standard Error of Mean 0.073
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.27, 97.5% CI 2-sided [-0.44 to -0.10], Standard Error of Mean 0.076

51. Secondary Outcome: Change From Baseline to Month 6 in Mean Pain Score of DYSP
Description: The DYSP pain scale ranged from 0 (absent) to 3 (severe).
Time Frame: Baseline, Month 6 of Treatment Period
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 203 | 149 | 120
units on a scale | -0.29 (0.048) | -0.41 (0.057) | -0.60 (0.062)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.118, mixed-effects model; LS Mean of Difference = -0.12, 97.5% CI 2-sided [-0.28 to 0.05], Standard Error of Mean 0.074
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.30, 97.5% CI 2-sided [-0.48 to -0.13], Standard Error of Mean 0.078

52. Secondary Outcome: Change From Baseline to Month 1 in Analgesic Use Across Both Classes of Rescue Analgesics
Description: as for outcome 6
Time Frame: Baseline, Month 1 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: pills
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 372 | 248 | 245
pills | -0.20 (0.028) | -0.25 (0.034) | -0.32 (0.034)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.313, mixed-effects model; LS Mean of Difference = -0.04, 97.5% CI 2-sided [-0.14 to 0.05], Standard Error of Mean 0.044
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p = 0.006, mixed-effects model; LS Mean of Difference = -0.12, 97.5% CI 2-sided [-0.22 to -0.02], Standard Error of Mean 0.044

53. Secondary Outcome: Change From Baseline to Month 2 in Analgesic Use Across Both Classes of Rescue Analgesics
Description: as for outcome 6
Time Frame: Baseline, Month 2 of Treatment Period
Population: The modified intent-to-treat analysis set included all randomized participants who took at least 1 dose of randomized, double-blind study drug. Observed cases.
Measure: Least Squares Mean (Standard Error); unit: pills
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 348 | 232 | 221
pills | -0.24 (0.029) | -0.27 (0.036) | -0.46 (0.037)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.519, mixed-effects model; LS Mean of Difference = -0.03, 97.5% CI 2-sided [-0.13 to 0.07], Standard Error of Mean 0.047
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.22, 97.5% CI 2-sided [-0.32 to -0.11], Standard Error of Mean 0.047

54. Secondary Outcome: Change From Baseline to Month 4 in Analgesic Use Across Both Classes of Rescue Analgesics
Description: as for outcome 7
Time Frame: Baseline, Month 4 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: pills
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 316 | 219 | 198
pills | -0.28 (0.033) | -0.39 (0.041) | -0.57 (0.042)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.037, mixed-effects model; LS Mean of Difference = -0.11, 97.5% CI 2-sided [-0.23 to 0.01], Standard Error of Mean 0.053
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.29, 97.5% CI 2-sided [-0.41 to -0.17], Standard Error of Mean 0.053

55. Secondary Outcome: Change From Baseline to Month 5 in Analgesic Use Across Both Classes of Rescue Analgesics
Description: as for outcome 6
Time Frame: Baseline, Month 5 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: pills
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 299 | 202 | 191
pills | -0.29 (0.034) | -0.36 (0.041) | -0.60 (0.042)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.200, mixed-effects model; LS Mean of Difference = -0.07, 97.5% CI 2-sided [-0.19 to 0.05], Standard Error of Mean 0.053
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.30, 97.5% CI 2-sided [-0.42 to -0.18], Standard Error of Mean 0.054

56. Secondary Outcome: Response to Patient Global Impression of Change (PGIC) at Month 1
Description: The PGIC questionnaire is a self-reported 7-point scale rating a participant's overall impression of change from 1 = very much improved to 7 = very much worse. Participants evaluated the change in their endometriosis-associated pain since initiation of study drug.
Time Frame: Month 1 of Treatment Period
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 353 | 234 | 226
units on a scale | 3.50 (0.060) | 2.97 (0.073) | 2.76 (0.075)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -0.53, 95% CI 2-sided [-0.72 to -0.34], Standard Error of Mean 0.094
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -0.74, 95% CI 2-sided [-0.93 to -0.56], Standard Error of Mean 0.095

57. Secondary Outcome: Response to PGIC at Month 2
Description: as for outcome 56
Time Frame: Month 2 of Treatment Period
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 353 | 231 | 225
units on a scale | 3.13 (0.062) | 2.74 (0.076) | 2.11 (0.077)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -0.39, 95% CI 2-sided [-0.58 to -0.19], Standard Error of Mean 0.098
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -1.02, 95% CI 2-sided [-1.21 to -0.82], Standard Error of Mean 0.099

58. Secondary Outcome: Response to PGIC at Month 3
Description: as for outcome 56
Time Frame: Month 3 of Treatment Period
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 346 | 229 | 227
units on a scale | 3.14 (0.064) | 2.53 (0.079) | 2.01 (0.079)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -0.61, 95% CI 2-sided [-0.81 to -0.41], Standard Error of Mean 0.101
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -1.12, 95% CI 2-sided [-1.32 to -0.92], Standard Error of Mean 0.102

59. Secondary Outcome: Response to PGIC at Month 4
Description: as for outcome 56
Time Frame: Month 4 of Treatment Period
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 352 | 230 | 222
units on a scale | 3.16 (0.067) | 2.54 (0.082) | 1.91 (0.084)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -0.63, 95% CI 2-sided [-0.83 to -0.42], Standard Error of Mean 0.106
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -1.26, 95% CI 2-sided [-1.47 to -1.05], Standard Error of Mean 0.107

60. Secondary Outcome: Response to PGIC at Month 5
Description: as for outcome 56
Time Frame: Month 5 of Treatment Period
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 350 | 233 | 223
units on a scale | 3.19 (0.070) | 2.50 (0.086) | 1.87 (0.088)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -0.69, 95% CI 2-sided [-0.91 to -0.48], Standard Error of Mean 0.111
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -1.32, 95% CI 2-sided [-1.54 to -1.10], Standard Error of Mean 0.112

61. Secondary Outcome: Response to PGIC at Month 6
Description: as for outcome 56
Time Frame: Month 6 of Treatment Period
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 308 | 207 | 200
units on a scale | 3.27 (0.077) | 2.56 (0.094) | 1.92 (0.096)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -0.72, 95% CI 2-sided [-0.96 to -0.48], Standard Error of Mean 0.122
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANOVA; LS Mean of Difference = -1.35, 95% CI 2-sided [-1.59 to -1.11], Standard Error of Mean 0.123

62. Secondary Outcome: Change From Baseline to Month 1 in NRS Scores
Description: The NRS for overall endometriosis-associated pain ranges 0 (none) to 10 (worst pain ever).
Time Frame: Baseline, Month 1 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 372 | 248 | 244
units on a scale | -0.72 (0.069) | -1.00 (0.085) | -1.12 (0.085)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.011, mixed-effects model; LS Mean of Difference = -0.28, 95% CI 2-sided [-0.52 to -0.03], Standard Error of Mean 0.109
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.40, 97.5% CI 2-sided [-0.65 to -0.16], Standard Error of Mean 0.110

63. Secondary Outcome: Change From Baseline to Month 2 in NRS Scores
Description: The NRS for overall endometriosis-associated pain ranges 0 (none) to 10 (worst pain ever).
Time Frame: Baseline, Month 2 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 348 | 232 | 221
units on a scale | -0.91 (0.086) | -1.38 (0.106) | -1.87 (0.107)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.47, 97.5% CI 2-sided [-0.77 to -0.16], Standard Error of Mean 0.137
Statistical Analysis 2: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = -0.96, mixed-effects model; LS Mean of Difference = -0.96, 97.5% CI 2-sided [-1.27 to -0.65], Standard Error of Mean 0.138

64. Secondary Outcome: Change From Baseline to Month 4 in NRS Scores
Description: The NRS for overall endometriosis-associated pain ranges 0 (none) to 10 (worst pain ever).
Time Frame: Baseline, Month 4 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 316 | 219 | 198
units on a scale | -1.15 (0.103) | -1.95 (0.126) | -2.76 (0.129)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.80, 97.5% CI 2-sided [-1.17 to -0.44], Standard Error of Mean 0.163
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -1.61, 97.5% CI 2-sided [-1.98 to -1.24], Standard Error of Mean 0.165

65. Secondary Outcome: Change From Baseline to Month 5 in NRS Scores
Description: The NRS for overall endometriosis-associated pain ranges 0 (none) to 10 (worst pain ever).
Time Frame: Baseline, Month 5 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 299 | 202 | 191
units on a scale | -1.24 (0.106) | -1.92 (0.129) | -2.85 (0.132)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.68, 97.5% CI 2-sided [-1.05 to -0.30], Standard Error of Mean 0.167
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -1.61, 97.5% CI 2-sided [-1.99 to -1.23], Standard Error of Mean 0.170

66. Secondary Outcome: Change From Baseline to Month 6 in NRS Scores
Description: The NRS for overall endometriosis-associated pain ranges 0 (none) to 10 (worst pain ever).
Time Frame: Baseline, Month 6 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 288 | 198 | 182
units on a scale | -1.15 (0.112) | -1.80 (0.136) | -2.75 (0.140)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -0.65, 97.5% CI 2-sided [-1.04 to -0.25], Standard Error of Mean 0.176
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, mixed-effects model; LS Mean of Difference = -1.60, 97.5% CI 2-sided [-2.00 to -1.20], Standard Error of Mean 0.179

67. Secondary Outcome: Change From Baseline to Month 1 in the Pain Domain of the Endometriosis Health Profile-30 (EHP-30)
Description: The EHP-30 is a disease-specific self-administered questionnaire used to measure health-related quality of life in women with endometriosis. Each domain is calculated on a scale from 0 = best possible health status to 100 = worst possible health status.
Time Frame: Baseline, Month 1 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 345 | 233 | 217
units on a scale | -14.47 (0.997) | -20.76 (1.213) | -24.23 (1.257)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -6.29, 95% CI 2-sided [-9.37 to -3.21], Standard Error of Mean 1.57
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -9.76, 95% CI 2-sided [-12.91 to -6.61], Standard Error of Mean 1.60

68. Secondary Outcome: Change From Baseline to Month 3 in the Pain Domain of the EHP-30
Description: as for outcome 67
Time Frame: Baseline, Month 3 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 312 | 217 | 197
units on a scale | -17.71 (1.101) | -26.99 (1.321) | -36.46 (1.386)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -9.28, 95% CI 2-sided [-12.66 to -5.91], Standard Error of Mean 1.72
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -18.75, 95% CI 2-sided [-22.22 to -15.27], Standard Error of Mean 1.77

69. Secondary Outcome: Change From Baseline to Month 6 in the Pain Domain of the EHP-30
Description: The EHP-30 is a disease-specific self-administered questionnaire used to measure health-related quality of life in women with endometriosis. Each domian is calculated on a scale from 0 = best possible health status to 100 = worst possible health status.
Time Frame: Baseline, Month 6 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 249 | 177 | 162
units on a scale | -15.42 (1.283) | -27.99 (1.522) | -40.52 (1.591)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -12.57, 95% CI 2-sided [-16.48 to -8.66], Standard Error of Mean 1.99
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -25.10, 95% CI 2-sided [-29.12 to -21.09], Standard Error of Mean 2.04

70. Secondary Outcome: Change From Baseline to Month 1 in the Sexual Intercourse Domain of the EHP-30
Description: as for outcome 69
Time Frame: Baseline, Month 1 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 248 | 172 | 146
units on a scale | -10.47 (1.239) | -11.26 (1.488) | -15.52 (1.614)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.685, ANCOVA; LS Mean of Difference = -0.78, 95% CI 2-sided [-4.59 to 3.02], Standard Error of Mean 1.94
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p = 0.013, ANCOVA; Difference in LS Means = -5.04, 95% CI 2-sided [-9.04 to -1.05], Standard Error of Mean 2.03

71. Secondary Outcome: Change From Baseline to Month 3 in the Sexual Intercourse Domain of the EHP-30
Description: as for outcome 67
Time Frame: Baseline, Month 3 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 228 | 167 | 133
units on a scale | -12.57 (1.551) | -17.32 (1.813) | -26.44 (2.032)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.047, ANCOVA; Difference in LS Means = -4.74, 95% CI 2-sided [-9.43 to -0.05], Standard Error of Mean 2.39
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -13.86, 95% CI 2-sided [-18.89 to -8.84], Standard Error of Mean 2.56

72. Secondary Outcome: Change From Baseline to Month 6 in the Sexual Intercourse Domain of the EHP-30
Description: as for outcome 69
Time Frame: Baseline, Month 6 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 170 | 128 | 110
units on a scale | -11.56 (1.909) | -16.27 (2.203) | -29.07 (2.384)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.107, ANCOVA; Difference in LS Means = -4.71, 95% CI 2-sided [-10.43 to 1.02], Standard Error of Mean 2.91
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -17.51, 95% CI 2-sided [-23.52 to -11.50], Standard Error of Mean 3.06

73. Secondary Outcome: Change From Baseline to Month 1 in Health Related Productivity Questionnaire (HRPQ): Number of Hours of Work Lost From Workplace Due to Absenteeism
Description: The HRPQ consists of questions measuring the impact of endometriosis-associated pain and its treatment on work productivity (number of work hours lost from the workplace due to absenteeism) in the 7 days prior to survey administration.
Time Frame: Baseline, Month 1 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 251 | 171 | 162
hours | -1.32 (0.236) | -1.20 (0.286) | -2.49 (0.294)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.741, ANCOVA; Difference in LS Means = 0.12, 95% CI 2-sided [-0.61 to 0.85], Standard Error of Mean 0.37
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p = 0.002, ANCOVA; Difference in LS Means = -1.16, 95% CI 2-sided [-1.90 to -0.42], Standard Error of Mean 0.38

74. Secondary Outcome: Change From Baseline to Month 2 in HRPQ: Number of Hours of Work Lost From Workplace Due to Absenteeism
Description: as for outcome 73
Time Frame: Baseline, Month 2 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 232 | 160 | 147
hours | -1.29 (0.222) | -1.77 (0.266) | -2.56 (0.278)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.172, ANCOVA; Difference in LS Means = -0.47, 95% CI 2-sided [-1.16 to 0.21], Standard Error of Mean 0.35
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -1.27, 95% CI 2-sided [-1.97 to -0.57], Standard Error of Mean 0.36

75. Secondary Outcome: Change From Baseline to Month 3 in HRPQ: Number of Hours of Work Lost From Workplace Due to Absenteeism
Description: as for outcome 73
Time Frame: Baseline, Month 3 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 215 | 148 | 140
hours | -0.87 (0.277) | -1.92 (0.333) | -2.65 (0.343)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.016, ANCOVA; LS Mean of Difference = -1.05, 95% CI 2-sided [-1.90 to -0.19], Standard Error of Mean 0.43
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -1.78, 95% CI 2-sided [-2.65 to -0.91], Standard Error of Mean 0.44

76. Secondary Outcome: Change From Baseline to Month 4 in HRPQ: Number of Hours of Work Lost From Workplace Due to Absenteeism
Description: as for outcome 73
Time Frame: Baseline, Month 4 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 205 | 148 | 134
hours | -1.08 (0.284) | -1.85 (0.334) | -2.44 (0.351)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.080, ANCOVA; Difference in LS Means = -0.77, 95% CI 2-sided [-1.63 to 0.09], Standard Error of Mean 0.44
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p = 0.003, ANCOVA; Difference in LS Means = -1.37, 95% CI 2-sided [-2.25 to -0.48], Standard Error of Mean 0.45

77. Secondary Outcome: Change From Baseline to Month 5 in HRPQ: Number of Hours of Work Lost From Workplace Due to Absenteeism
Description: as for outcome 73
Time Frame: Baseline, Month 5 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 209 | 147 | 128
hours | -1.10 (0.258) | -1.75 (0.308) | -2.94 (0.330)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.106, ANCOVA; Difference in LS Means = -0.65, 95% CI 2-sided [-1.44 to 0.14], Standard Error of Mean 0.40
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -1.85, 95% CI 2-sided [-2.67 to -1.02], Standard Error of Mean 0.42

78. Secondary Outcome: Change From Baseline to Month 6 in HRPQ: Number of Hours of Work Lost From Workplace Due to Absenteeism
Description: as for outcome 73
Time Frame: Baseline, Month 6 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 159 | 120 | 105
hours | -0.27 (0.409) | -1.02 (0.471) | -2.48 (0.503)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.232, ANCOVA; Difference in LS Means = -0.75, 95% CI 2-sided [-1.97 to 0.48], Standard Error of Mean 0.62
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -2.21, 95% CI 2-sided [-3.48 to -0.93], Standard Error of Mean 0.65

79. Secondary Outcome: Change From Baseline to Month 1 in HRPQ: Number of Hours of Work Lost From Household Due to Absenteeism
Description: The HRPQ consists of questions measuring the impact of endometriosis-associated pain and its treatment on work productivity (number of work hours lost from the household due to absenteeism) in the 7 days prior to survey administration.
Time Frame: Baseline, Month 1 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 319 | 200 | 202
hours | -1.27 (0.229) | -2.19 (0.289) | -2.89 (0.288)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.013, ANCOVA; Difference in LS Means = -0.92, 95% CI 2-sided [-1.65 to -0.20], Standard Error of Mean 0.37
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -1.62, 95% CI 2-sided [-2.35 to -0.90], Standard Error of Mean 0.37

80. Secondary Outcome: Change From Baseline to Month 2 in HRPQ: Number of Hours of Work Lost From Household Due to Absenteeism
Description: as for outcome 79
Time Frame: Baseline, Month 2 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 287 | 192 | 183
hours | -1.43 (0.295) | -2.75 (0.360) | -3.06 (0.369)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.005, ANCOVA; Difference in LS Means = -1.33, 95% CI 2-sided [-2.24 to -0.41], Standard Error of Mean 0.47
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -1.64, 95% CI 2-sided [-2.56 to -0.71], Standard Error of Mean 0.47

81. Secondary Outcome: Change From Baseline to Month 3 in HRPQ: Number of Hours of Work Lost From Household Due to Absenteeism
Description: as for outcome 79
Time Frame: Baseline, Month 3 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 278 | 185 | 179
hours | -1.37 (0.292) | -3.00 (0.358) | -3.47 (0.363)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -1.63, 95% CI 2-sided [-2.53 to -0.72], Standard Error of Mean 0.46
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -2.10, 95% CI 2-sided [-3.02 to -1.19], Standard Error of Mean 0.47

82. Secondary Outcome: Change From Baseline to Month 4 in HRPQ: Number of Hours of Work Lost From Household Due to Absenteeism
Description: as for outcome 79
Time Frame: Baseline, Month 4 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 264 | 170 | 171
hours | -1.38 (0.265) | -2.59 (0.331) | -3.61 (0.330)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.004, ANCOVA; Difference in LS Means = -1.21, 95% CI 2-sided [-2.05 to -0.38], Standard Error of Mean 0.42
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -2.23, 95% CI 2-sided [-3.06 to -1.40], Standard Error of Mean 0.42

83. Secondary Outcome: Change From Baseline to Month 5 in HRPQ: Number of Hours of Work Lost From Household Due to Absenteeism
Description: as for outcome 79
Time Frame: Baseline, Month 5 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 253 | 173 | 171
hours | -2.13 (0.250) | -3.10 (0.302) | -3.94 (0.304)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.013, ANCOVA; Difference in LS Means = -0.97, 95% CI 2-sided [-1.74 to -0.20], Standard Error of Mean 0.39
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -1.81, 95% CI 2-sided [-2.58 to -1.04], Standard Error of Mean 0.39

84. Secondary Outcome: Change From Baseline to Month 6 in HRPQ: Number of Hours of Work Lost From Household Due to Absenteeism
Description: as for outcome 79
Time Frame: Baseline, Month 6 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 191 | 145 | 139
hours | -1.45 (0.313) | -2.73 (0.359) | -3.94 (0.367)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.007, ANCOVA; Difference in LS Means = -1.28, 95% CI 2-sided [-2.22 to -0.34], Standard Error of Mean 0.48
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -2.49, 95% CI 2-sided [-3.44 to -1.54], Standard Error of Mean 0.48

85. Secondary Outcome: Change From Baseline to Month 1 in HRPQ: Number of Hours of Work Lost From Workplace Due to Presenteeism
Description: The HRPQ consists of questions measuring the impact of endometriosis-associated pain and its treatment on work productivity (number of work hours lost from the workplace due to presenteeism [working while sick]) in the 7 days prior to survey administration.
Time Frame: Baseline, Month 1 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 246 | 170 | 157
hours | -4.07 (0.555) | -4.93 (0.668) | -6.00 (0.694)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.326, ANCOVA; Difference in LS Means = -0.86, 95% CI 2-sided [-2.57 to 0.85], Standard Error of Mean 0.87
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p = 0.031, ANCOVA; Difference in LS Means = -1.93, 95% CI 2-sided [-3.67 to -0.18], Standard Error of Mean 0.89

86. Secondary Outcome: Change From Baseline to Month 2 in HRPQ: Number of Hours of Work Lost From Workplace Due to Presenteeism
Description: as for outcome 85
Time Frame: Baseline, Month 2 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 228 | 158 | 145
hours | -5.42 (0.560) | -6.83 (0.671) | -8.94 (0.701)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.107, ANCOVA; Difference in LS Means = -1.41, 95% CI 2-sided [-3.13 to 0.31], Standard Error of Mean 0.88
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -3.52, 95% CI 2-sided [-5.28 to -1.75], Standard Error of Mean 0.90

87. Secondary Outcome: Change From Baseline to Month 3 in HRPQ: Number of Hours of Work Lost From Workplace Due to Presenteeism
Description: as for outcome 85
Time Frame: Baseline, Month 3 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 213 | 147 | 136
hours | -6.23 (0.526) | -7.24 (0.632) | -9.16 (0.657)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.219, ANCOVA; Difference in LS Means = -1.01, 95% CI 2-sided [-2.63 to 0.60], Standard Error of Mean 0.82
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -2.93, 95% CI 2-sided [-4.59 to -1.28], Standard Error of Mean 0.84

88. Secondary Outcome: Change From Baseline to Month 4 in HRPQ: Number of Hours of Work Lost From Workplace Due to Presenteeism
Description: as for outcome 85
Time Frame: Baseline, Month 4 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 201 | 146 | 132
hours | -6.81 (0.465) | -8.41 (0.546) | -10.70 (0.573)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.026, ANCOVA; Difference in LS Means = -1.60, 95% CI 2-sided [-3.01 to -0.19], Standard Error of Mean 0.72
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -3.89, 95% CI 2-sided [-5.34 to -2.43], Standard Error of Mean 0.74

89. Secondary Outcome: Change From Baseline to Month 5 in HRPQ: Number of Hours of Work Lost From Workplace Due to Presenteeism
Description: as for outcome 85
Time Frame: Baseline, Month 5 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 206 | 147 | 123
hours | -7.80 (0.488) | -8.31 (0.577) | -10.93 (0.631)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.502, ANCOVA; Difference in LS Means = -0.51, 95% CI 2-sided [-2.00 to 0.98], Standard Error of Mean 0.76
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -3.13, 95% CI 2-sided [-4.70 to -1.56], Standard Error of Mean 0.80

90. Secondary Outcome: Change From Baseline to Month 6 in HRPQ: Number of Hours of Work Lost From Workplace Due to Presenteeism
Description: as for outcome 85
Time Frame: Baseline, Month 6 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 157 | 118 | 104
hours | -6.75 (0.554) | -8.11 (0.637) | -11.21 (0.679)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.108, ANCOVA; Difference in LS Means = -1.36, 95% CI 2-sided [-3.02 to 0.30], Standard Error of Mean 0.85
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -4.47, 95% CI 2-sided [-6.19 to -2.74], Standard Error of Mean 0.88

91. Secondary Outcome: Change From Baseline to Month 1 in HRPQ: Number of Hours of Work Lost From Household Due to Presenteeism
Description: The HRPQ consists of questions measuring the impact of endometriosis-associated pain and its treatment on work productivity (number of work hours lost from the household due to presenteeism [working while sick]) in the 7 days prior to survey administration.
Time Frame: Baseline, Month 1 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 314 | 200 | 199
hours | -0.46 (0.224) | -1.64 (0.281) | -1.51 (0.282)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.001, ANCOVA; Difference in LS Means = -1.19, 95% CI 2-sided [-1.90 to -0.48], Standard Error of Mean 0.36
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p = 0.004, ANCOVA; Difference in LS Means = -1.05, 95% CI 2-sided [-1.76 to -0.34], Standard Error of Mean 0.36

92. Secondary Outcome: Change From Baseline to Month 2 in HRPQ: Number of Hours of Work Lost From Household Due to Presenteeism
Description: as for outcome 91
Time Frame: Baseline, Month 2 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 285 | 190 | 181
hours | -1.17 (0.238) | -1.93 (0.291) | -2.23 (0.299)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.045, mixed-effects model; Difference in LS Means = -0.76, 95% CI 2-sided [-1.49 to -0.02], Standard Error of Mean 0.38
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p = 0.006, ANCOVA; Difference in LS Means = -1.06, 95% CI 2-sided [-1.81 to -0.31], Standard Error of Mean 0.38

93. Secondary Outcome: Change From Baseline to Month 3 in HRPQ: Number of Hours of Work Lost From Household Due to Presenteeism
Description: as for outcome 91
Time Frame: Baseline, Month 3 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 275 | 185 | 178
hours | -1.35 (0.210) | -1.89 (0.256) | -2.33 (0.261)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.103, ANCOVA; Difference in LS Means = -0.54, 95% CI 2-sided [-1.19 to 0.11], Standard Error of Mean 0.33
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p = 0.003, ANCOVA; Difference in LS Means = -0.98, 95% CI 2-sided [-1.64 to -0.32], Standard Error of Mean 0.34

94. Secondary Outcome: Change From Baseline to Month 4 in HRPQ: Number of Hours of Work Lost From Household Due to Presenteeism
Description: as for outcome 91
Time Frame: Baseline, Month 4 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 263 | 168 | 170
hours | -1.51 (0.224) | -1.81 (0.280) | -2.55 (0.278)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.390, ANCOVA; Difference in LS Means = -0.31, 95% CI 2-sided [-1.01 to 0.40], Standard Error of Mean 0.36
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p = 0.003, ANCOVA; Difference in LS Means = -1.05, 95% CI 2-sided [-1.75 to -0.35], Standard Error of Mean 0.36

95. Secondary Outcome: Change From Baseline to Month 5 in HRPQ: Number of Hours of Work Lost From Household Due to Presenteeism
Description: as for outcome 91
Time Frame: Baseline, Month 5 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 253 | 172 | 169
hours | -1.67 (0.169) | -1.86 (0.205) | -2.71 (0.206)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.460, ANCOVA; Difference in LS Means = -0.20, 95% CI 2-sided [-0.72 to 0.32], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -1.04, 95% CI 2-sided [-1.57 to -0.52], Standard Error of Mean 0.27

96. Secondary Outcome: Change From Baseline to Month 6 in HRPQ: Number of Hours of Work Lost From Household Due to Presenteeism
Description: as for outcome 91
Time Frame: Baseline, Month 6 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 191 | 145 | 135
hours | -1.48 (0.232) | -2.07 (0.265) | -2.78 (0.275)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.095, ANCOVA; LS Mean of Difference = -0.59, 95% CI 2-sided [-1.28 to 0.10], Standard Error of Mean 0.35
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -1.30, 95% CI 2-sided [-2.01 to -0.59], Standard Error of Mean 0.36

97. Secondary Outcome: Change From Baseline to Month 1 in HRPQ: Total (Absenteeism and Presenteeism) Number of Hours of Work Lost From Workplace
Description: The HRPQ consists of questions measuring the impact of endometriosis-associated pain and its treatment on work productivity (number of work hours lost from the workplace due to absenteeism and presenteeism) in the 7 days prior to survey administration.
Time Frame: Baseline, Month 1 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 251 | 171 | 162
hours | -5.46 (0.615) | -6.17 (0.745) | -8.69 (0.764)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.462, ANCOVA; Difference in LS Means = -0.71, 95% CI 2-sided [-2.61 to 1.19], Standard Error of Mean 0.97
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p = 0.001, ANCOVA; Difference in LS Means = -3.23, 95% CI 2-sided [-5.16 to -1.30], Standard Error of Mean 0.98

98. Secondary Outcome: Change From Baseline to Month 2 in HRPQ: Total (Absenteeism and Presenteeism) Number of Hours of Work Lost From Workplace
Description: as for outcome 97
Time Frame: Baseline, Month 2 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 232 | 160 | 147
hours | -6.70 (0.621) | -8.72 (0.746) | -11.56 (0.778)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.039, ANCOVA; Difference in LS Means = -2.02, 95% CI 2-sided [-3.93 to -0.11], Standard Error of Mean 0.97
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -4.86, 95% CI 2-sided [-6.82 to -2.90], Standard Error of Mean 1.00

99. Secondary Outcome: Change From Baseline to Month 3 in HRPQ: Total (Absenteeism and Presenteeism) Number of Hours of Work Lost From Workplace
Description: as for outcome 97
Time Frame: Baseline, Month 3 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 215 | 148 | 140
hours | -7.00 (0.654) | -9.20 (0.787) | -11.90 (0.808)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.032, ANCOVA; Difference in LS Means = -2.20, 95% CI 2-sided [-4.21 to -0.18], Standard Error of Mean 1.03
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -4.91, 95% CI 2-sided [-6.95 to -2.86], Standard Error of Mean 1.04

100. Secondary Outcome: Change From Baseline to Month 4 in HRPQ: Total (Absenteeism and Presenteeism) Number of Hours of Work Lost From Workplace
Description: as for outcome 97
Time Frame: Baseline, Month 4 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 205 | 148 | 134
hours | -7.84 (0.605) | -10.26 (0.712) | -13.09 (0.747)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.010, ANCOVA; Difference in LS Means = -2.42, 95% CI 2-sided [-4.26 to -0.58], Standard Error of Mean 0.94
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -5.25, 95% CI 2-sided [-7.14 to -3.36], Standard Error of Mean 0.96

101. Secondary Outcome: Change From Baseline to Month 5 in HRPQ: Total (Absenteeism and Presenteeism) Number of Hours of Work Lost From Workplace
Description: as for outcome 97
Time Frame: Baseline, Month 5 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 209 | 147 | 128
hours | -8.87 (0.604) | -10.04 (0.719) | -14.00 (0.771)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.215, ANCOVA; Difference in LS Means = -1.17, 95% CI 2-sided [-3.02 to 0.68], Standard Error of Mean 0.94
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -5.13, 95% CI 2-sided [-7.06 to -3.20], Standard Error of Mean 0.98

102. Secondary Outcome: Change From Baseline to Month 6 in HRPQ: Total (Absenteeism and Presenteeism) Number of Hours of Work Lost From Workplace
Description: as for outcome 97
Time Frame: Baseline, Month 6 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 159 | 120 | 105
hours | -6.88 (0.761) | -9.14 (0.874) | -13.67 (0.936)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.053, ANCOVA; Difference in LS Means = -2.25, 95% CI 2-sided [-4.53 to 0.03], Standard Error of Mean 1.16
Statistical Analysis 2: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -6.79, 95% CI 2-sided [-9.17 to -4.41], Standard Error of Mean 1.21

103. Secondary Outcome: Change From Baseline to Month 1 in HRPQ: Total (Absenteeism and Presenteeism) Number of Hours of Work Lost From Household
Description: The HRPQ consists of questions measuring the impact of endometriosis-associated pain and its treatment on work productivity (number of work hours lost from the household due to absenteeism and presenteeism) in the 7 days prior to survey administration.
Time Frame: Baseline, Month 1 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 319 | 200 | 202
hours | -1.76 (0.352) | -3.88 (0.445) | -4.36 (0.443)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -2.12, 95% CI 2-sided [-3.24 to -1.01], Standard Error of Mean 0.57
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -2.60, 95% CI 2-sided [-3.71 to -1.49], Standard Error of Mean 0.57

104. Secondary Outcome: Change From Baseline to Month 2 in HRPQ: Total (Absenteeism and Presenteeism) Number of Hours of Work Lost From Household
Description: as for outcome 103
Time Frame: Baseline, Month 2 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 287 | 192 | 183
hours | -2.60 (0.423) | -4.69 (0.517) | -5.25 (0.529)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.002, ANCOVA; Difference in LS Means = -2.09, 95% CI 2-sided [-3.40 to -0.78], Standard Error of Mean 0.67
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -2.65, 95% CI 2-sided [-3.98 to -1.32], Standard Error of Mean 0.68

105. Secondary Outcome: Change From Baseline to Month 3 in HRPQ: Total (Absenteeism and Presenteeism) Number of Hours of Work Lost From Household
Description: as for outcome 103
Time Frame: Baseline, Month 3 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 278 | 185 | 179
hours | -2.73 (0.394) | -4.90 (0.483) | -5.73 (0.492)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -2.17, 95% CI 2-sided [-3.39 to -0.95], Standard Error of Mean 0.62
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -3.00, 95% CI 2-sided [-4.23 to -1.76], Standard Error of Mean 0.63

106. Secondary Outcome: Change From Baseline to Month 4 in HRPQ: Total (Absenteeism and Presenteeism) Number of Hours of Work Lost From Household
Description: as for outcome 103
Time Frame: Baseline, Month 4 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 264 | 170 | 171
hours | -2.89 (0.403) | -4.43 (0.502) | -6.13 (0.501)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.017, ANCOVA; Difference in LS Means = -1.54, 95% CI 2-sided [-2.80 to -0.27], Standard Error of Mean 0.64
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -3.24, 95% CI 2-sided [-4.50 to -1.98], Standard Error of Mean 0.64

107. Secondary Outcome: Change From Baseline to Month 5 in HRPQ: Total (Absenteeism and Presenteeism) Number of Hours of Work Lost From Household
Description: as for outcome 103
Time Frame: Baseline, Month 5 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 253 | 173 | 171
hours | -3.80 (0.349) | -4.94 (0.423) | -6.62 (0.425)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.038, ANCOVA; Difference in LS Means = -1.14, 95% CI 2-sided [-2.22 to -0.07], Standard Error of Mean 0.55
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -2.83, 95% CI 2-sided [-3.91 to -1.74], Standard Error of Mean 0.55

108. Secondary Outcome: Change From Baseline to Month 6 in HRPQ: Total (Absenteeism and Presenteeism) Number of Hours of Work Lost From Household
Description: as for outcome 103
Time Frame: Baseline, Month 6 of Treatment Period
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 191 | 145 | 139
hours | -2.94 (0.433) | -4.78 (0.496) | -6.69 (0.507)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg QD; Test type: Superiority; p = 0.006, ANCOVA; Difference in LS Means = -1.83, 95% CI 2-sided [-3.13 to -0.54], Standard Error of Mean 0.66
Statistical Analysis 2: Comparison: Placebo vs Elagolix 200 mg BID; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS Means = -3.75, 95% CI 2-sided [-5.06 to -2.44], Standard Error of Mean 0.67

109. Secondary Outcome: Number of Participants With Endometriosis-Related Non-Study Health Visits During the Treatment Period
Time Frame: Up to Month 6 of Treatment Period
Population: The modified intent-to-treat analysis set included all randomized participants who took at least 1 dose of randomized, double-blind study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 374 | 249 | 248
Participants
  Baseline | 69 | 54 | 51
  Month 1 | 70 | 50 | 47
  Month 2 | 59 | 38 | 33
  Month 3 | 66 | 37 | 48
  Month 4 | 54 | 35 | 42
  Month 5 | 43 | 32 | 22
  Month 6 | 38 | 26 | 21
  Overall | 189 | 126 | 113

110. Secondary Outcome: Number of Days of Hospitalization
Time Frame: Up to Month 6 of Treatment Period
Population: The modified intent-to-treat analysis set included all randomized participants who took at least 1 dose of randomized, double-blind study drug. Includes participants who were hospitalized during the Treatment Period.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 15 | 3 | 13
days | 2.9 (2.45) | 2.0 (1.00) | 2.0 (1.68)

111. Secondary Outcome: Number of Participants With Emergency Room/Outpatient Procedures During the Treatment Period, by Type
Time Frame: Up to Month 6 of Treatment Period
Population: as for outcome 109
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Elagolix 150 mg QD | Elagolix 200 mg BID
Number analyzed (Participants) | 374 | 249 | 248
Participants
  All Categories | 62 | 21 | 32
  Abdominal Hysterectomy | 0 | 0 | 0
  Angiography | 0 | 0 | 0
  Arthroscopy | 0 | 0 | 1
  Biopsy | 1 | 0 | 1
  Blood Draw | 27 | 7 | 16
  Consultation | 6 | 3 | 3
  CT Scan | 21 | 3 | 6
  Diagnostic Laparoscopy | 0 | 1 | 0
  Electrocardiogram | 3 | 1 | 3
  Endometrial Ablation | 0 | 0 | 0
  Histological Exam | 0 | 0 | 0
  Intrauterine Insemination | 0 | 0 | 0
  In Vitro Fertilization | 0 | 0 | 0
  Laparoscopic Hysterectomy | 0 | 0 | 0
  Laparotomy | 0 | 0 | 0
  Magnetic Resonance Imaging | 0 | 0 | 0
  Oophorectomy | 0 | 0 | 0
  Pelvic Exam | 5 | 1 | 2
  Physical Examination | 32 | 10 | 15
  Surgery for Adhesions | 0 | 0 | 0
  Therapeutic Laparoscopy | 0 | 0 | 1
  Transfusion | 0 | 0 | 0
  Ultrasound | 14 | 3 | 6
  Urine Test | 26 | 8 | 11
  Vaginal Hysterectomy | 0 | 0 | 0
  X-Ray | 14 | 2 | 5
  Other (Not Specified) | 16 | 10 | 10

ADVERSE EVENTS:
Time Frame: From first dose of study treatment through 6 months of treatment plus up to 12 months of follow-up.
Description: Adverse events (AEs) are defined as treatment-emergent if they began on or after the date of the first dose of study drug through up to 30 days after the last dose of study drug for participants who did not enroll in the separate extension study (Study M12-667, NCT01760954). For participants who enrolled in the separate extension study, treatment-emergent AEs are those that began on or after the first dose of study drug until the day prior to the first dose date in the extension study.
Arm/Group | Placebo | Elagolix 150 MG QD | Elagolix 200 MG BID
Serious Adverse Events (participants affected / at risk) | 12/374 | 2/249 | 7/248
Other Adverse Events (participants affected / at risk) | 180/374 | 147/249 | 159/248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=374) | Elagolix 150 MG QD (N=249) | Elagolix 200 MG BID (N=248)
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 0
CHEST PAIN (General disorders) | 1 | 1 | 0
APPENDICITIS (Infections and infestations) | 1 | 0 | 1
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 | 0 | 0
MENINGITIS VIRAL (Infections and infestations) | 1 | 0 | 0
PYELONEPHRITIS (Infections and infestations) | 0 | 0 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
BLOOD POTASSIUM DECREASED (Investigations) | 1 | 0 | 0
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
ECTOPIC PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
ANXIETY (Psychiatric disorders) | 0 | 0 | 1
CALCULUS URETERIC (Renal and urinary disorders) | 0 | 0 | 1
HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 0 | 1
URETERIC STENOSIS (Renal and urinary disorders) | 0 | 1 | 0
ENDOMETRIOSIS (Reproductive system and breast disorders) | 1 | 0 | 2
HAEMORRHAGIC OVARIAN CYST (Reproductive system and breast disorders) | 1 | 0 | 0
OVARIAN CYST RUPTURED (Reproductive system and breast disorders) | 0 | 0 | 1
PELVIC PAIN (Reproductive system and breast disorders) | 1 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
VICTIM OF SEXUAL ABUSE (Social circumstances) | 1 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=374) | Elagolix 150 MG QD (N=249) | Elagolix 200 MG BID (N=248)
NAUSEA (Gastrointestinal disorders) | 51 | 25 | 40
VOMITING (Gastrointestinal disorders) | 19 | 11 | 10
FATIGUE (General disorders) | 23 | 14 | 16
NASOPHARYNGITIS (Infections and infestations) | 7 | 13 | 11
SINUSITIS (Infections and infestations) | 17 | 14 | 12
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 24 | 19 | 8
URINARY TRACT INFECTION (Infections and infestations) | 36 | 19 | 16
BACK PAIN (Musculoskeletal and connective tissue disorders) | 26 | 10 | 10
HEADACHE (Nervous system disorders) | 37 | 38 | 43
ANXIETY (Psychiatric disorders) | 15 | 6 | 15
DEPRESSION (Psychiatric disorders) | 10 | 9 | 13
INSOMNIA (Psychiatric disorders) | 9 | 16 | 18
AMENORRHOEA (Reproductive system and breast disorders) | 1 | 8 | 14
ACNE (Skin and subcutaneous tissue disorders) | 16 | 13 | 10
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 5 | 6 | 14
HOT FLUSH (Vascular disorders) | 26 | 59 | 105

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.